CLINICAL TRIAL: NCT04061551
Title: Eliminate Hepatitis C/EC Partnership Evaluation Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: Burnet Institute (Other); The Alfred (Other); St Vincent's Hospital Melbourne (Other); HepatitisVictoria (Unknown); Harm Reduction Australia (Unknown); Victoria State Government (Unknown); Gilead Sciences (Industry); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HREC/16/Alfred/164
Record Dates: First submitted 2019-06-04; First posted 2019-08-20 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis C; Chronic Hepatitis c; Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Intervention Model Description: The comprehensive intervention will be implemented at all participating sites, although specific components of the intervention will be tailored to the needs of each site. The model consists of five stages:
  1. Baseline site assessment
  2. Co-design intervention to streamline HCV clinical pathways
  3. Implementation
  4. Six-monthly review
  5. End line review
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EC Clinic Support (Experimental): Whole of practice interventions delivery through nurse-led model
  Interventions: Other: EC clinic support - whole of practice interventions delivery through nurse-led model

INTERVENTIONS:
Other: EC clinic support - whole of practice interventions delivery through nurse-led model — The primary interventions will be delivered through a team of nurses, an evaluation team and practice support team that will be working with each of the services to improved Hepatitis C service delivery.
  The EC project team will predominantly be involved in working with providers and staff at EC sites to implement key interventions that have been collated into a Primary Care Practice Toolkit, which cover three domains; patient support, provider support and practice Support. The toolkit is designed to be an educational and implementation resource that the nursing team will support services to deliver.
  * Patient support to reduce the impact of hepatitis C and other blood borne viruses
  * Provider support to reduce the impact of hepatitis C and other blood borne viruses
  * Practice support to reduce the impact of hepatitis C and other blood borne viruses

SUMMARY:
The Eliminate Hepatitis C (EC) Partnership project is a multi-site, multi-year project aiming to enhance and extend hepatitis C virus (HCV) care and treatment among people who inject drugs (PWID) through nurse-led models of care in the community and the prison system. The project will implement and evaluate a health service intervention to enhance HCV response by improving health promotion, offering training and education to service providers, streamlining clinical pathways, utilising data systems and surveillance and implementing the results of ongoing research and evaluation.

Health services data will be used to assess the impact of the EC nurse-led support, to enhance the clinical pathway and increase HCV testing, linkage to care and treatment uptake in community and prison settings. This will include provider and client interviews and a sentinel surveillance system (ACCESS) that will track and monitor impact indicators including HCV testing, linkage to care and treatment uptake at the service and population level.

Overall, evaluation data will be used to monitor the uptake of HCV treatment in PWID, monitor the effectiveness of community- and prison-based treatment program and assess the cost and feasibility of treating >1160 PWID in community-/prison-based program and assess changes in HCV prevalence in Victoria and modelling the impact of treating PWID to inform HCV elimination models in Australia and globally.

DETAILED DESCRIPTION:
An estimated 71 million people are living with hepatitis C virus (HCV) world-wide, at significant risk of morbidity and mortality from liver cirrhosis, liver failure and hepatocellular carcinoma. However, the development of well-tolerated, highly-efficacious curative direct-acting antiviral treatment (DAAs) has contributed to a global push to eliminate HCV as a public health threat. The World Health Organization has developed a global strategy for elimination that calls for 90% of people living with HCV to be diagnosed and 90% of those diagnosed to be treated by 2030.

In 2015, prior to the DAAs being released, it was estimated that around 230,000 people living with HCV in Australia. Like in many other high-income countries, the group most affected by HCV in Australia are people who inject drugs (PWID), making this a key population group for Australia's HCV elimination efforts.

Despite the availability of DAAs through Australia's Pharmaceutical Benefits Scheme (PBS), numerous barriers exist for PWID to access HCV care and particularly to accessing tertiary-based care. As such, targeting community-based services that provide comprehensive care packages for PWID, including the provision of opioid substitution therapy (OST), counselling, a needle and syringe program (NSP) for the delivery of HCV treatment should increase PWIDs' engagement in HCV care. The EC Partnership program has been funded to increase capacity of community and prison services to provide HCV testing and treatment with DAA treatments by streamlining clinical pathways and reducing barriers to access.

The EC Partnership project is a multi-site, multi-year project aiming to enhance and extend hepatitis C virus (HCV) care and treatment among people who inject drugs (PWID) through nurse-led models of care in the community and the prison system. Specifically the project aims to:

* Increase demand for HCV treatment among PWID;
* Increase the capacity of community services to provide HCV testing & treatment with PBS listed DAAs;
* Increase the capacity to provide HCV testing & treatment in prison with PBS listed DAAs;
* Streamline clinical pathways (tailored for different types of settings) to increase access to PBS listed DAAs; and
* Establish an integrated HCV surveillance system to more accurately monitor trends in HCV prevalence and incidence over time.

To achieve this, the project will implement and evaluate a health service intervention for prison-based and community-based health services providing care to PWID. The intervention will have five main components:

1. enhance HCV response by improving health promotion;
2. offering training and education to service providers;
3. streamlining clinical pathways;
4. utilising data systems and surveillance;
5. and implementing the results of ongoing research and evaluation.

The intervention will be evaluated using qualitative and quantitative data from health services, clinical providers and clients, which will include:

* EC experience observational cohort data will assess predictors of patient engagement and identify barriers and enablers to progression through the cascade of care
* Interviews with clinical service providers to assess changes to clinical pathways and to inform cost-effectiveness analysis
* Clinical data from the Australian Collaboration for Co-ordinated Sentinel Surveillance (ACCESS) System that will track and monitor impact indictors including HCV testing, linkage to care and treatment uptake at the service and population level
* Data from State-wide Hepatitis Assessment and Management Program (Prison programs)
* Data from Medicare, PBS and other Victorian Department of Health and Human Services datasets (This will occur with a subset of patients who provide consent from participating sites).

In addition, the project will incorporate a sub study (Ophelia evaluation) that will be used to guide development and implementation of health promotion initiatives.

The EC Partnership evaluation aims to measure the overall impact of the EC Partnership by monitoring and evaluating specific key outcomes, including:

* Number of PWID who uptake HCV treatment across EC partnerships services within the community and the prison system;
* Treatment effectiveness (SVR12 cure rates & treatment failures) among community and the prison based treatment programs, compared to tertiary-based treatment programs;
* Cost and feasibility of treating >1,160 PWID within the community and the prison systems;
* Changes in HCV prevalence and incidence in Victoria, and comparing community and prison population estimates;
* Model the impact of treating PWID to inform HCV elimination models in Australia and globally.

ELIGIBILITY:
The level of recruitment is clinics rather than individuals. Eligible clinics are those with a high HCV caseload, with a focus on drug and alcohol community clinics and general practitioners.

Eligibility criteria for individuals providing information in the form of interviews will be:

* 18 years of age or older; AND
* Willing and able to provide informed, written consent to participate; AND
* Either of:

  * staff of a participating EC site who are involved in hepatitis C care; OR
  * clients of a participating EC site who attend the site for screening and management of hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of treatment amongst PWID | 5 years
  The number of PWID who commence HCV treatment across EC partnerships sites over time and compared to tertiary care models

SECONDARY OUTCOMES:
Treatment effectiveness relative to tertiary care services | 5 years
  Rates of cure, assessed as sustained virological response at 12 weeks post treatment completion (SVR12), and treatment failure amongst PWID treatment in community and prison-based services will be compared to tertiary-based treatment programs.
Costs of scaling up treatment for PWID | 5 years
  The costs of treating >1,160 PWID within the community and prison services will be assessed.
Changes in HCV prevalence and incidence in Victoria | 5 years
  HCV prevalence and incidence will be tracked during the project and compared to historical data.
Projected impact on HCV elimination targets | 5 years
  Mathematical modelling studies will assess the expected impact the changes in treatment uptake, incidence and prevalence will have on the WHO incidence and mortality targets for viral hepatitis elimination. This will be used to provide an estimate of the feasibility of achieving elimination targets in Australia and in other countries.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret E Hellard, MD PhD, Principal Investigator — Burnet Institute and Alfred Health
Locations (1):
- Burnet Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scott N, McBryde ES, Thompson A, Doyle JS, Hellard ME. Treatment scale-up to achieve global HCV incidence and mortality elimination targets: a cost-effectiveness model. Gut. 2017 Aug;66(8):1507-1515. doi: 10.1136/gutjnl-2016-311504. Epub 2016 Apr 12. PMID 27196586
- [Background] Scott N, Doyle JS, Wilson DP, Wade A, Howell J, Pedrana A, Thompson A, Hellard ME. Reaching hepatitis C virus elimination targets requires health system interventions to enhance the care cascade. Int J Drug Policy. 2017 Sep;47:107-116. doi: 10.1016/j.drugpo.2017.07.006. Epub 2017 Aug 7. PMID 28797497
- [Background] Doyle JS, Scott N, Sacks-Davis R, Pedrana AE, Thompson AJ, Hellard ME; Eliminate Hepatitis C Partnership. Treatment access is only the first step to hepatitis C elimination: experience of universal anti-viral treatment access in Australia. Aliment Pharmacol Ther. 2019 May;49(9):1223-1229. doi: 10.1111/apt.15210. Epub 2019 Mar 25. PMID 30908706